CLINICAL TRIAL: NCT00964912
Title: Placebo-Controlled, Ascending Single-Dose Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of BMS-820836 in Healthy Subjects
Brief Title: Single Dose Study of BMS-820836
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CN162-001
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — 6-(2-methyl-4-(2-naphthyl)-1,2,3,4-tetrahydroisoquinolin-7-yl)pyridazin-3-amine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (11):
- BMS-820836 (Part 1, Panel 1) (Active Comparator)
  Interventions: Drug: BMS-820836; Drug: Placebo
- BMS-820836 (Part 1, Panel 2) (Active Comparator)
  Interventions: Drug: BMS-820836; Drug: Placebo
- BMS-820836 (Part 1, Panel 3) (Active Comparator)
  Interventions: Drug: BMS-820836; Drug: Placebo
- BMS-820836 (Part 1, Panel 4) (Active Comparator)
  Interventions: Drug: BMS-820836; Drug: Placebo
- BMS-820836 (Part 1, Panel 5) (Active Comparator)
  Interventions: Drug: BMS-820836; Drug: Placebo
- BMS-820836 (Part 1, Panel 6) (Active Comparator)
  Interventions: Drug: BMS-820836; Drug: Placebo
- BMS-820836 (Part 1, Panel 7) (Active Comparator)
  Interventions: Drug: BMS-820836; Drug: Placebo
- BMS-820836 (Part 1, Panel 8) (Active Comparator)
  Interventions: Drug: BMS-820836; Drug: Placebo
- BMS-820836 (Part 1, Panel 9) (Active Comparator)
  Interventions: Drug: BMS-820836; Drug: Placebo
- BMS-820836 (Part 2, Panel A) (Active Comparator)
  Interventions: Drug: BMS-820836
- BMS-820836 (Part 2, Panel B) (Active Comparator)
  Interventions: Drug: BMS-820836

INTERVENTIONS:
Drug: BMS-820836 — Oral Solution, Oral, 0.025 mg, single dose, one dose
  Arms: BMS-820836 (Part 1, Panel 1)
Drug: BMS-820836 — Oral Solution, Oral, 0.1 mg, single dose, one dose
  Arms: BMS-820836 (Part 1, Panel 2)
Drug: BMS-820836 — Oral Solution, Oral, 0.25 mg, single dose, one dose
  Arms: BMS-820836 (Part 1, Panel 3)
Drug: BMS-820836 — Oral Solution, Oral, 0.5 mg, single dose, one dose
  Arms: BMS-820836 (Part 1, Panel 4)
Drug: BMS-820836 — Oral Solution, Oral, 1 mg, single dose, one dose
  Arms: BMS-820836 (Part 1, Panel 5)
Drug: BMS-820836 — Oral Solution, Oral, 2 mg, single dose, one dose
  Arms: BMS-820836 (Part 1, Panel 6)
Drug: BMS-820836 — Oral Solution, Oral, 3 mg, single dose, one dose
  Arms: BMS-820836 (Part 1, Panel 7)
Drug: BMS-820836 — Oral Solution, Oral, 5 mg, single dose, one dose
  Arms: BMS-820836 (Part 1, Panel 8)
Drug: BMS-820836 — Oral Solution, Oral, 8 mg, single dose, one dose
  Arms: BMS-820836 (Part 1, Panel 9)
Drug: Placebo — Oral Solution, Oral, 0 mg, single dose, one dose
  Arms: BMS-820836 (Part 1, Panel 1); BMS-820836 (Part 1, Panel 2); BMS-820836 (Part 1, Panel 3); BMS-820836 (Part 1, Panel 4); BMS-820836 (Part 1, Panel 5); BMS-820836 (Part 1, Panel 6); BMS-820836 (Part 1, Panel 7); BMS-820836 (Part 1, Panel 8); BMS-820836 (Part 1, Panel 9)
Drug: BMS-820836 — Oral Solution, Oral, 3 mg, single dose, one dose
  Arms: BMS-820836 (Part 2, Panel A)
Drug: BMS-820836 — Oral Solution, Oral, 0.5 mg, single dose, one dose
  Arms: BMS-820836 (Part 2, Panel B)

SUMMARY:
The purpose of this study is to determine the safety and tolerability of BMS-820836 after single doses

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 18 to 30 kg/m2, inclusive and weight ≥ 50 kg
* Right-handed, non-ambidextrous subjects for Part 2
* Men and women, ages 18 to 55 years, inclusive

Exclusion Criteria:

* Women of child bearing potential (WOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 8 weeks after the last dose of investigational product
* WOCBP using a prohibited contraceptive method
* Women who are pregnant or breastfeeding
* Sexually active fertile men not using effective birth control if their partners are WOCBP
* Any significant acute or chronic medical illness
* Current or recent (within 3 months) gastrointestinal disease
* History of cholecystectomy
* Any major surgery within 4 weeks of study drug administration
* Any gastrointestinal surgery that could impact the absorption of study drug
* Donation of blood or plasma to a blood bank or in a clinical study (except a screening visit) within 4 weeks of study drug administration
* Blood transfusion within 4 weeks of study drug administration
* Inability to tolerate/swallow oral medication
* Difficulty with venipuncture and/or poor venous access
* Self-reported smokers
* Recent (within 1 year) of psychostimulant use (cocaine, methylphenidate, amphetamines, ecstasy)
* Confirmed resting supine systolic blood pressure > 130 mmHg
* Confirmed resting supine diastolic blood pressure > 80 mmHg
* Confirmed QT value ≥ 500 msec
* Confirmed QTc (Bazett) value ≥ 450 msec
* History of any significant drug allergy (such as anaphylaxis or hepatotoxicity)
* History of peppermint allergies
* History of brain conditions (e.g. history of stroke, head trauma, etc.)
* History of or current psychiatric conditions
* History of claustrophobia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of BMS-820836 following single-dose administration | Within 14 days of first dose

SECONDARY OUTCOMES:
To assess the single-dose pharmacokinetics of BMS-820836 and its N-demethylated metabolite BMS-821007 | Within 7 days of dosing
To assess the pharmacodynamics of BMS-820836 | Within 48 hours of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Toronto, Ontario, Canada

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx